CLINICAL TRIAL: NCT02211014
Title: An Open-Label, Phase 1b Study of ACP-196 With and Without Dexamethasone in Subjects With Multiple Myeloma
Brief Title: An Open-Label, Phase 1b Study of Acalabrutinib With and Without Dexamethasone in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Collaborators: Acerta Pharma, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACE-MY-001
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma (MM)
Keywords: Bruton tyrosine kinase inhibitor; Btk; Multiple Myeloma; MM; ACP-196; acalabrutinib; Calquence
MeSH Terms: conditions — Multiple Myeloma | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Acalabrutinib 100 mg twice daily (bid) continuously
  Interventions: Drug: acalabrutinib
- Cohort 2 (Experimental): Acalabrutinib 100 mg bid continuously and 40 mg dexamethasone once weekly
  Interventions: Drug: acalabrutinib

INTERVENTIONS:
Drug: acalabrutinib
  Other Names: ACP-196

SUMMARY:
To characterize the safety profile of acalabrutinib with and without dexamethasone in subjects with relapsed or refractory Multiple Myeloma (MM)

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* A confirmed diagnosis of MM, which has relapsed after, or been refractory to ≥ 1 prior therapy for MM, and is progressing at the time of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Agreement to use contraception during the study and for 30 days after the last dose of study drugs if sexually active and able to bear or beget children.

Exclusion Criteria:

* A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk
* Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, gastric bypass, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
* Breast feeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613
Locations (3):
- Baltimore, Maryland, United States
- United Kingdom (2):
  - United Kingdom, Leicester
  - Guys and St Thomas' Hospital NHS Foundation Trust, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter, open-label, randomized, parallel-group study to evaluate the safety, pharmacokinetics, pharmacodynamics and activity of acalabrutinib with/without dexamethasone in subjects with relapsed/refractory multiple myeloma in US and United Kingdom. 27 subjects enrolled into 2 cohorts. Enrollment was discontinued because of lack of efficacy.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 13 | 14
Completed | 11 | 8
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Started another cancer therapy | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — In agreement with patient, no benefit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 4 | 13
  >=65 years | 4 | 10 | 14
Age, Continuous [Median (Full Range); unit: years] | 60.0 [49 to 83] | 68.5 [53 to 78] | 65.0 [49 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 14 | 25
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 7 | 13
  United Kingdom | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of Acalabrutinib With and Without Dexamethasone
Description: AEs and SAEs were coded by system organ class (SOC) and preferred term (PT) based on the Medical Dictionary for Regulatory Activities (MedDRA) reporting system. All AEs summarized were treatment-emergent. Summaries were also presented by the severity of the AE (per Common Toxicity Criteria for Adverse Events [CTCAE]) and by relationship to study drug as assessed by the investigator. Events of clinical interest (ECIs) selected for dedicated analysis were evaluated using Standardized MedDRA Queries, where available, by SOC, or by Sponsor-defined baskets of MedDRA Adverse Event Grouped Terms (AEGTs). The following ECIs were summarized: Cardiac events (including a subset of atrial fibrillation), cytopenias (anemia, leukopenia, neutropenia, and thrombocytopenia), hemorrhage (including a subset of major hemorrhage), hepatic events, hypertension, infection, interstitial lung disease/pneumonitis, second primary malignancies (second primary malignancies excluding skin), tumor lysis syndrome.
Time Frame: From first dose of study drug up to Cycle 12 (48 weeks). Subjects who showed benefit from study drugs were allowed to continue until disease progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 13 | 14
Participants
  Treatment-emergent adverse events (TEAE) | 13 | 14
  Treatment-related TEAE | 7 | 7
  SAE | 5 | 9
  Treatment-related SAE | 1 | 2
  TEAE leading to actions taken on study drug | 1 | 8

2. Secondary Outcome: Pharmacokinetic (PK) Parameters Calculated for Acalabrutinib: AUC0-4, AUClast, AUCINF, Cmax, Tmax, λz, t1/2, CL/F, and Vz/F. PK Parameters Calculated for Dexamethasone: Tmax, Cmax, AUC0-4 and AUClast.
Description: The plasma PK of study drug was characterized using noncompartmental analysis. PK parameters were calculated whenever possible, from plasma concentrations of acalabrutinib. Missing dates or times could have been imputed for PK and pharmacodynamic (PD) samples if the missing values could be established with an acceptable level of accuracy based on other information obtained during the visit in question. If PK and PD sampling for a 33 Final Clinical Study Report Drug Substance Acalabrutinib Study Code ACE-MY-001 Edition Number 2 Date 31 October 2018 given subject was not performed according to protocol, the subject could have been excluded from the PK and PD analyses. The PK parameters were tabulated and summarized using descriptive statistics. For each PD variable, the concentration at each assessment was described. The change from baseline to each assessment was summarized. As appropriate the on treatment values were compared with the pretreatment baseline values using paired t-tests.
Time Frame: On Days 1 and 22: pre-dose, and at 0.5, 0.75, 1, 2, 4, and 6 hours after the morning dose. On Days 8, 15, and 28: pre-dose and 1 hour after the morning dose.
Population: Day 1: 24 (of 27 subjects enrolled) were equally randomized (1:1 ratio) into two cohorts to receive Acalabrutinib (12 in Cohort 1), or with dexamethasone (12 in Cohort 2).
  Day 22: 17 (of 24) subjects with PK data were remaining: 9 in Cohort 1 and 8 in Cohort 2. Seven subjects discontinued the study prior to Day 22.
Measure: Mean (Standard Deviation); unit: percentage of CV
Groups:
- Cohort 1 - Day 1; Cohort 1 - Day 22: Acalabrutinib 100 mg twice daily (bid) continuously
- Cohort 2 - Day 1; Cohort 2 - Day 22: Acalabrutinib 100 mg bid continuously and 40 mg dexamethasone once weekly
Arm/Group | Cohort 1 - Day 1 | Cohort 2 - Day 1 | Cohort 1 - Day 22 | Cohort 2 - Day 22
Number analyzed (Participants) | 12 | 12 | 9 | 8
percentage of CV
  Cmax (ng/mL) - the maximum concentration observed | 524 (112) | 437 (91.5) | 271 (103) | 607 (90.8)
  AUC (area under the curve)_0-4 (hr*ng/mL) | 604 (72.9) | 621 (64) | 390 (105) | 766 (60.5)
  AUC_last (hr*ng/mL) | 638 (69.5) | 675 (56.9) | 423 (102) | 812 (58.3)
  AUC_INF (infinity) (hr*ng/mL) | 754 (67.8) | 732 (63.1) | 411 (111) | 826 (62.6)

3. Secondary Outcome: Bruton Tyrosine Kinase (BTK) Occupancy
Description: The percent occupied BTK was calculated in each subject's peripheral blood mononuclear cells (PBMC) sample for each assessment timepoint using an ELISA-based method. Samples from 17 subjects met the criteria for data inclusion, having a dynamic range (signal to noise) of ≥5 for the Day 1 pre-dose timepoint. Acalabrutinib administered at 100 mg bid resulted in a median steady-state (Day 8) BTK target occupancy level of 95% and 98% for Cohort 1 and Cohort 2, respectively. The Days 28 and 56 assessments, both taken at pre-dose, were >97% occupancy for each cohort. Intersubject variability was low, with 6 of 7 (86%) subjects in Cohort 1 and 4 of 5 (80%) subjects in Cohort 2 having >90% BTK occupancy at steady-state trough (12h post-dose). The single subject in Cohort 2 with <90% occupancy at Day 8 pre-dose did not take their Day 7 doses.
Time Frame: On Days 1 and 8: pre-dose and at 4 hours after the morning dose. On Days 28 and 56: morning pre-dose only.
Population: 17 (of 27) subjects with evaluable data. For 10 subjects the data was excluded due to: no Day 1 sample received, low cells events or parent populations, or other deviation.
  Day 1 post and additional time points, further decrease of evaluable data due to: subject discontinuation, low cells events or parent populations, or other deviation.
Measure: Mean (Standard Deviation); unit: percentage of occupied BTK
Groups:
- Cohort 1 - Day 1 Pre; Cohort 1 - Day 1 Post; Cohort 1 - Day 8 Pre; Cohort 1 - Day 8 Post; Cohort 1 - Day 28 Pre; Cohort 1 - Day 56 Pre: Acalabrutinib 100 mg twice daily (bid) continuously
- Cohort 2 - Day 1 Pre; Cohort 2 - Day 1 Post; Cohort 2 - Day 8 Pre; Cohort 2 - Day 8 Post; Cohort 2 - Day 28 Pre; Cohort 2 - Day 56 Pre: Acalabrutinib 100 mg bid continuously and 40 mg dexamethasone once weekly
Arm/Group | Cohort 1 - Day 1 Pre | Cohort 2 - Day 1 Pre | Cohort 1 - Day 1 Post | Cohort 2 - Day 1 Post | Cohort 1 - Day 8 Pre | Cohort 2 - Day 8 Pre | Cohort 1 - Day 8 Post | Cohort 2 - Day 8 Post | Cohort 1 - Day 28 Pre | Cohort 2 - Day 28 Pre | Cohort 1 - Day 56 Pre | Cohort 2 - Day 56 Pre
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 7 | 5 | 7 | 6 | 7 | 6 | 5 | 4
percentage of occupied BTK | 0 (0) | 0 (0) | 98.5 (0.9) | 98.5 (1.3) | 93.2 (6.6) | 94.3 (8.8) | 98.6 (1.1) | 96.8 (4.8) | 97.6 (1.8) | 95.8 (5.5) | 95.7 (6.2) | 97.6 (1.3)

4. Secondary Outcome: Response Assessed According to Guidelines Proposed by the International Myeloma Workshop Consensus Panel and European Group for Blood and Marrow Transplant
Description: Per EBMT: CR, negative immunofixation of serum and urine, disappearance of plasmacytomas and < 5% plasma cells; Stringent complete response (SCR), CR + normal flow cytometry and absence of clonal plasma cells; Very good partial response (VGPR), Serum and urine M-protein detectable on immunofixation but not on electrophoresis or > 90% reduction is serum and urine M protein; Partial response (PR), > 50% reduction in serum M-protein and > 90% reduction in 24 hour urine M-protein, > 50% reduction in baseline soft tissue plasmacytoma; Minimal response (MR), 25-49% reduction of serum M-protein and 50-59% reduction in 24 hour urine M-protein, 25-49% reduction in plasmacytomas and no increase in lytic bone lesions; Stable disease (SD), not meeting criteria for CR, VGPR, MR, PR or progressive disease (PD); PD, increase of 25% or more from nadir in serum M-protein, urine M-protein, new or increased bone lesions or plasmacytomas, or hypercalcemia solely attributed to multiple myeloma.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 13 | 14
Participants
  sCR | 0 | 0
  CR | 0 | 0
  VGPR | 0 | 0
  PR | 0 | 0
  MR | 1 | 2
  SD | 5 | 6
  PD | 4 | 1
  NE (not evaluable) | 3 | 5

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Day 0 and on or before Day 1210.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 2/13 | 4/14
Serious Adverse Events (participants affected / at risk) | 5/13 | 9/14
Other Adverse Events (participants affected / at risk) | 13/13 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2 (N=14)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Norovirus test positive (Investigations) | 0 | 1
Pain (General disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Renail impairment (Renal and urinary disorders) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2 (N=14)
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Headache (Nervous system disorders) | 6 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Fatigue (General disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Confusional state (Psychiatric disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Contusion (Psychiatric disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Pyrexia (General disorders) | 0 | 2
Rhinitis (Infections and infestations) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Cardiac murmur (Investigations) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 2 | 0
Platelet count decreased (Investigations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site and PI can publish/publicly present the results of the study only with prior written consent of Sponsor or otherwise after expiry of 12 months following completion of the study.

Site and PI agree to provide 30 days written notice to Sponsor prior to submission for publication or presentation."

DOCUMENTS (2):
  • Study Protocol (2016-01-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT02211014/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/14/NCT02211014/SAP_001.pdf